CLINICAL TRIAL: NCT00736060
Title: Study the Clinical and Laboratory Characteristics and the Outcome of Sickle Cell Anemia Patients Admitted to the Pediatric Ward Because of Fever as the Presenting Symptom
Brief Title: Clinical and Laboratory Characteristics of Sickle Cell Anemia Patients Admitted With Fever
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0027-08-EMC
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Sickle Cell Anemia; Sickle Cell Thalassemia
Keywords: Fever; Blood cultures
MeSH Terms: conditions — Anemia, Sickle Cell; Fever | interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Sickle cell anemia
  Interventions: Other: Observational
- 2: Sickle cell thalassemia
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Summary of clinical and laboratory data

SUMMARY:
This study will summarized the clinical and laboratory data and the outcome of all the patients suffering from Sickle Cell Anemia (Including Sickle cell thalassemia) admitted to the pediatric ward.

DETAILED DESCRIPTION:
The actual protocol for SCA patients admitted with fever is to obtain blood cultures and start empiric antibiotic treatment.

The study cohort included 60 SCA patients actually treated in the Pediatric Hematology Unit.

ELIGIBILITY:
Inclusion Criteria: All patients admitted with fever as the only presenting symptom.

Exclusion Criteria: Patients admitted with another causes related or unrelated to sickle cell disease and have also fever.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 patients treated at the Pediatric Hematology Unit in the Ha'Emek Medical Center suffering from sickle cell anemia or sickle cell thalassemia admitted with fever as the presenting symptom.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carina Levin, MD, Principal Investigator — Pediatric Hematology Unit - Ha'Emek Medical Center - Afula - 18101 - Israel; Ilena Arshinov, MD, Principal Investigator — Pediatric Dpt B - Ha'Emek Medical Center - Afula - Israel
Locations (1):
- Pediatric Hematology Unit - Ha'Emek Medical Center, Afula, Afula, Israel